CLINICAL TRIAL: NCT07111754
Title: How Can Behavioural Intent to Take Antibiotics "Exactly as Prescribed" be Increased? An Online Randomised Behavioural Experiment
Brief Title: Testing Interventions Designed to Improve How Members of the General Public Follow Instructions to Take Antibiotics
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: The Behavioural Insights Team (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 7836387
Record Dates: First submitted 2025-07-17; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Antibiotic Use
Keywords: Antibiotics; Behaviour Change; Randomised controlled trial; Antibiotic Resistance; Antimicrobial Resistance

STUDY DESIGN:
Intervention Model Description: The study intervention aims to change behavioural intent regarding the use of antibiotics. It is a 7 armed parallel randomised controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Control (No Intervention): Control arm, with a picture of a typical antibiotic packet shown to participants
- Behavioural Message - QR code (Experimental): Antibiotic packet with a QR code as the mechanism of delivery of the intervention, the intervention only contains information about the desired behaviour
  Interventions: Behavioral: Behavioural Message
- Behavioural Message - Warning (Experimental): Antibiotic packet with a warning message on it as the mechanism of delivery of the intervention, the intervention only contains information about the desired behaviour
  Interventions: Behavioral: Behavioural Message
- Behavioural message + positive framing - QR code (Experimental): Antibiotic packet with a QR code as the mechanism of delivery of the intervention, the intervention contains information about the desired behaviour and antimicrobial resistance (framed in a positive manner)
  Interventions: Behavioral: Behavioural message + positive framing
- Behavioural message + positive framing - Warning (Experimental): Antibiotic packet with a warning message on it as the mechanism of delivery of the intervention, the intervention contains information about the desired behaviour and antimicrobial resistance (framed in a positive manner)
  Interventions: Behavioral: Behavioural message + positive framing
- Behavioural message + negative framing - QR Code (Experimental): Antibiotic packet with a QR code as the mechanism of delivery of the intervention, the intervention contains information about the desired behaviour and antimicrobial resistance (framed in a negative manner)
  Interventions: Behavioral: Behavioural message + negative framing
- Behavioural message + negative framing - Warning (Experimental): Antibiotic packet with a warning message on it as the mechanism of delivery of the intervention, the intervention contains information about the desired behaviour and antimicrobial resistance (framed in a negative manner)
  Interventions: Behavioral: Behavioural message + negative framing

INTERVENTIONS:
Behavioral: Behavioural Message — Participants are presented with an image of an antibiotic packet, that contains information about the behaviour "take antibiotics exactly as prescribed". This can be delivered to participants via a QR code, or a warning message on the packet.
  Arms: Behavioural Message - QR code; Behavioural Message - Warning
Behavioral: Behavioural message + positive framing — Participants are presented with an image of an antibiotic packet, that contains information about the behaviour "take antibiotics exactly as prescribed" and information about AMR, framed in a positive manner. This can be delivered to participants via a QR code, or a warning message on the packet.
  Arms: Behavioural message + positive framing - QR code; Behavioural message + positive framing - Warning
Behavioral: Behavioural message + negative framing — Participants are presented with an image of an antibiotic packet, that contains information about the behaviour "take antibiotics exactly as prescribed" and information about AMR, framed in a negative manner. This can be delivered to participants via a QR code, or a warning message on the packet.
  Arms: Behavioural message + negative framing - QR Code; Behavioural message + negative framing - Warning

SUMMARY:
Antimicrobial resistance (AMR) is a global public health challenge. Due to overuse of antibiotics, bacteria are becoming resistant to antibiotics, which creates infections that can't be treated by modern medicine. To combat AMR, the public need to both know that AMR is an issue and know what actions they can take to address AMR.

When patients are prescribed antibiotics, the information provided (and how this is provided) is likely to be influential on whether they are taken correctly, or if behaviours that contribute to antimicrobial resistance (such as not finishing the course) predominate.

This study, a large online experiment involving 7,000 people across the UK, aims explore the influence of what information and how it is provided. The study looks at different ways of presenting information on antibiotic packets-from clear instructions to warnings and even scannable QR codes with extra details.

The main goals are to see if these changes can help participants understand how to take antibiotics exactly as prescribed. The investigators also want to see if it helps participants understand what antibiotic resistance is and their role in preventing it.

By understanding what works best, the investigators hope to find simple, effective ways to help everyone use antibiotics wisely, protecting these vital medicines for the future.

DETAILED DESCRIPTION:
Antimicrobial resistance (AMR), or antibiotic resistance, is a serious global health problem. It happens when bacteria evolve and become strong enough to resist the very antibiotics designed to kill them. This makes common infections much harder, or even impossible, to treat. A major reason for this growing threat is the overuse and misuse of antibiotics.

To fight AMR, it's crucial that the public not only understand that antibiotic resistance is a problem, but also know what steps can be taken to help. A key action is to take antibiotics exactly as prescribed. However, the investigators know that many people aren't entirely sure what "exactly as prescribed" really means. This can involve things like remembering to take the full course, taking it at the right times, and simply taking the medication at all.

To better understand these challenges, the Fleming Initiative conducted focus groups with the UK public in spring 2025. These discussions helped identify the main reasons people might not take antibiotics as directed, such as not understanding what "exactly as prescribed" means, or not knowing about AMR and how individual actions might contribute to it.

Using these insights, the Fleming Initiative then held co-design workshops with public participants. Together, several new ways to make it easier for individuals to take antibiotics correctly were developed.

This study is a seven-armed online behavioral experiment conducted in collaboration between the Fleming Initiative at Imperial College London, and the Behavioural Insights Team. It aims to understand how different presentations of information on antibiotic packaging about desired target behaviors and antimicrobial resistance (AMR) influence the public's correct antibiotic use, attitudes towards AMR, and future behavioral intent.

Primary Objective:

To measure the change in behavioral intent to "take antibiotics exactly as prescribed," using a composite measure of four individual behaviors related to antimicrobial stewardship (AMS).

Secondary Objectives:

To assess comprehension of how to take antibiotics. To assess comprehension of AMR.

Exploratory Objectives:

To evaluate changes in behavioral intent for individual behaviors related to "taking antibiotics exactly as prescribed" (e.g., finishing the course, number per day).

To understand if participants recognise that not taking antibiotics exactly as prescribed contributes to AMR.

To examine the impact of message framing and the mechanism of intervention delivery on behavioral intent to take antibiotics exactly as prescribed.

To assess the impact on perceived personal responsibility regarding AMR.

To determine the proportion of individuals who interacted with a QR code (in relevant arms).

To gauge the impact of interventions on sentiment towards information on the package itself.

To evaluate participants' opinions on whether text message reminders would help participants take antibiotics exactly as prescribed.

Study Design and Participant Recruitment:

The study will recruit 7,000 UK participants, aged 18 and over, through market research panels via the Predictiv online platform, an online survey platform created by the Behavioural Insights Team.

Participants will be randomised 1:1:1:1:1:1:1 into one of seven trial arms: a control arm with a standard antibiotic packet, and six intervention arms. Interventions include QR codes linking to additional information (Arms 2-4) and warning messages on the packaging (Arms 5-7).

Recruitment will use quotas for age, gender, region, and ethnicity to ensure a nationally representative sample.

The participant journey involves accessing the survey, an introduction slide, an attention check, randomisation, baseline measures of AMR understanding, a standardized medical scenario, exposure to their assigned antibiotic packet image (intervention), a series of survey questions, and finally, demographic questions.

Participants will be anonymous, with no personally identifying data transferred to the research team. Participants will receive a small financial incentive (£0.70) managed by the market research panels. The total study duration is anticipated to be around 3 weeks.

Sub-group Analysis:

The primary analysis will be repeated for subgroups based on age, health confidence, and baseline comprehension of AMR to identify differential impacts of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over
* United Kingdom residents
* Have passed the attention check at the start of the online survey.

Exclusion Criteria:

* Individuals who are not signed up a market research panel and therefore will not have access to the online survey.
* Those resident outside the UK.
* Those who fail the attention check at the start of the online survey. Individuals aged under 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7000 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2025-10-24 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall intent to take antibiotics as prescribed | During the intervention
  The proportion of Moderately, Very likely, or 'Yes' responses across the 4 measures of intent (taking one dose at a time, taking the full course, spacing the doses throughout the day, stopping when feeling better).

SECONDARY OUTCOMES:
Proportion of correct responses on comprehension questions about antibiotic use | During the intervention
  Responses to six questions relating to taking antibiotics exactly as prescribed, including how many per day, how many days for, when should tablets be taken, duration of course, how many tablets at a time and how to space across day

OTHER OUTCOMES:
Individual measures of intent to take antibiotics as prescribed | During the intervention
  Impact of intervention on individual behaviours relating to taking antibiotics as prescribed
Do the interventions increase understanding that not taking antibiotics as prescribed contributes to AMR? | During the intervention
What is the effect of changing the messaging of the intervention on overall intent to take antibiotics as prescribed | During the intervention
  Control vs Neutral framing vs positive framing vs negative framing
What is the effect of changing the mechanism of delivery of the intervention on overall intent to take antibiotics as prescribed | During the intervention
  Control vs QR code vs Warning message on packet
What is the effect of the intervention on personal responsibility? | During the intervention
  Personal responsibility associated with preventing AMR, according to behavioural intervention
Do the interventions change sentiment towards the information on the package itself? | During the intervention
  Total score for questions related to whether the information on the antibiotic packet was relevant to the participant

CONTACTS AND LOCATIONS:
Overall Officials: Kate Grailey, Principal Investigator — Imperial College London

IPD SHARING:
Plan to Share IPD: Yes
Anonymised participant data will be shared at the time of study publication on an openly available database

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT07111754/Prot_SAP_000.pdf